CLINICAL TRIAL: NCT05344118
Title: Parental Perceptions on Prescription Opioid Use for Pain Control in Children Undergoing Orthopedic Surgery
Brief Title: Parental Perceptions on Prescription Opioid Use
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Joseph D. Tobias, Chief of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Other Study IDs: STUDY00002410
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Results first posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parents: Parents of children undergoing orthopedic surgery
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — REDCap survey

SUMMARY:
This study involves an anonymous survey given to parents regarding their perceptions on prescription opioid use for pain control in children undergoing orthopedic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Parents of patients between 1-18 years of age scheduled for orthopedic surgery at Nationwide Children's Hospital.

Exclusion Criteria:

* Parents with children less than 1 or greater than 18 years of age or scheduled for surgery other than orthopedic.
* Non-English speaking parents.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Parents of children scheduled for orthopedic surgery
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Parents
Started | 125
Completed | 125
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Parents
Number analyzed (Participants) | 125
Age, Customized [Count of Participants; unit: Participants] — Population: Age data not collected via survey
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Sex/gender data not collected via survey
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 117
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 103
  More than one race | 3
  Unknown or Not Reported | 4
Relationship to child [Count of Participants; unit: Participants] — Population: 2 of the participants did not answer this question in the survey.
  Participants
    Father: number analyzed (Participants) | 123
    Father | 26
    Grandparent: number analyzed (Participants) | 123
    Grandparent | 5
    Legal Guardian: number analyzed (Participants) | 123
    Legal Guardian | 4
    Mother: number analyzed (Participants) | 123
    Mother | 88
Marital Status [Count of Participants; unit: Participants]
  Divorced or separated | 16
  Married or domestic partner | 81
  Single, never married | 25
  No answer | 3
Primary Language Spoken at Home [Count of Participants; unit: Participants]
  English | 118
  Other | 2
  No answer | 5

OUTCOME MEASURES:

1. Primary Outcome: Comfort With Child Receiving Opioids During Surgery
Description: Are you comfortable with your child receiving opioids (for example: Morphine, Fentanyl, Dilaudid) during surgery?
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Parents
Number analyzed (Participants) | 125
Participants
  No | 5
  Yes | 84
  Yes, but I have concerns | 36

2. Primary Outcome: Comfort With Child Receiving Opioids After Surgery
Description: Are you comfortable with your child receiving opioids (for example: Morphine, Fentanyl, Dilaudid) after surgery?
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Parents
Number analyzed (Participants) | 125
Participants
  No | 11
  Yes | 69
  Yes, but I have concerns | 45

3. Primary Outcome: Danger of Opioids
Description: Do you believe prescription opioids are dangerous?
Time Frame: Baseline
Population: Three of the 125 participants did not answer this question.
Measure: Count of Participants; unit: Participants
Arm/Group | Parents
Number analyzed (Participants) | 122
Participants
  No | 41
  Yes | 81

4. Primary Outcome: Opioid Education
Description: How much education have you received about opioids?
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Parents
Number analyzed (Participants) | 125
Participants
  None | 12
  Somewhat informed | 68
  Very informed | 45

5. Primary Outcome: Safe Storage of Opioids
Description: In your opinion, what is the most appropriate way to safely store opioids?
Time Frame: Baseline
Population: Three of the 125 participants did not answer this question.
Measure: Count of Participants; unit: Participants
Arm/Group | Parents
Number analyzed (Participants) | 122
Participants
  Don't know | 2
  In a locked place | 70
  Medicine cabinet | 5
  Out of reach of children | 45

6. Primary Outcome: Safe Disposal of Opioids
Description: In your opinion, what is the most appropriate way to safely dispose of opioids?
Time Frame: Baseline
Population: Two of the 125 participants did not answer this question.
Measure: Count of Participants; unit: Participants
Arm/Group | Parents
Number analyzed (Participants) | 123
Participants
  Don't know | 6
  Drop them in a disposal box | 25
  Flush them down the sink/disposal/toilet | 16
  Take them to a collection event | 30
  Take them to a pharmacy, doctor, or hospital | 45
  Throw them in the garbage | 1

7. Secondary Outcome: Employment Status
Description: Current employment status of parent
Time Frame: Baseline
Population: Three participants out of 125 did not answer this question.
Measure: Count of Participants; unit: Participants
Arm/Group | Parents
Number analyzed (Participants) | 122
Participants
  Employed for wages | 85
  Not working | 8
  Out of work and looking for work | 2
  Self-employed | 12
  Stay at home parent | 14
  Student | 1

8. Secondary Outcome: Education
Description: Level of education of parent
Time Frame: Baseline
Population: Four of the 125 participants did not answer this question.
Measure: Count of Participants; unit: Participants
Arm/Group | Parents
Number analyzed (Participants) | 121
Participants
  Advanced degree | 23
  Bachelor's degree | 16
  Between high school and college | 58
  High school graduate, diploma, or equivalent | 21
  Some high school, no diploma | 3

9. Secondary Outcome: Gender of Child
Description: Gender at birth of participant's child undergoing surgery
Time Frame: Baseline
Population: Two of the 125 participants did not answer this question.
Measure: Count of Participants; unit: Participants
Arm/Group | Parents
Number analyzed (Participants) | 123
Participants
  Female | 63
  Male | 60

10. Secondary Outcome: Age of Child
Description: Age of the participant's child undergoing surgery
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Parents
Number analyzed (Participants) | 125
years | 11.3 (4.2)

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Parents
All-Cause Mortality (participants affected / at risk) | 0/125
Serious Adverse Events (participants affected / at risk) | 0/125
Other Adverse Events (participants affected / at risk) | 0/125

LIMITATIONS AND CAVEATS:
The study had a relatively small sample size with limited heterogeneity of respondents which could have led to a lack of differences among specific demographic, educational, and socioeconomic groups. The study also limited enrollment to English speakers so that they could easily complete the survey on the iPad. As such, this may not be representative of the diversity that is present in our entire parent population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-12): https://cdn.clinicaltrials.gov/large-docs/18/NCT05344118/Prot_SAP_000.pdf